CLINICAL TRIAL: NCT05842330
Title: Benefits of In-prison OROS-methylphenidate vs. Placebo Treatment in Detained People With Attention-deficit/Hyperactivity Disorder: A Randomized Controlled Trial
Brief Title: Benefits of ADHD Treatment in Detained People
Acronym: BATIR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stéphanie Baggio (Other)
Collaborators: University of Lausanne (Other); University of Geneva, Switzerland (Other); Netherlands Institute for the Study of Crime (Unknown); School of Health Sciences Fribourg (Unknown)
Responsible Party: Sponsor-Investigator, Stéphanie Baggio, Prof., University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 32003B_212581
Record Dates: First submitted 2023-04-05; First posted 2023-05-06 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: ADHD
Keywords: Prison; Health care; Adherence to treatment; Recidivism
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Treatment Adherence and Compliance; Recidivism | interventions — Methylphenidate

STUDY DESIGN:
Intervention Model Description: This is a phase 3 parallel randomized controlled trial (1:1 ratio) of OROS-MPH vs. a placebo on a clinical outcome.
  Participants will undertake three months (12 weeks) of treatment while they are incarcerated. After three months, all participants will be offered treatment in outpatient care, either in prison or in the community. They will have daily monitoring of medical adherence in prison or in electronic monitors after release (without being unblinded on the treatment they received during detention). They will be followed-up for twelve months as outpatient care (total study duration: 15 months).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be blinded to the 3-month (12 weeks) in-prison treatment. The research team and statistician will be blinded to the participants' group. The psychiatrist will be unblinded when participants are released. At that time of the study, all participants will be offered to have the treatment (OROS-MPH) without being unblinded regarding their initial group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pharmaceutical intervention (OROS-MPH) (Experimental): Participants will receive OROS-MPH (Concerta® available in Switzerland as first-line treatment for ADHD). Dosages will be defined according to the Swiss Compendium. The psychiatrist (blinded during detention) will start with the smallest dosage (18 mg, Concerta®). The treatment will be monitored weekly the first month, and then monthly. The pharmacy of the Geneva University Hospitals will be in charge of over-encapsulating medications.
  Interventions: Drug: Concerta
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Concerta — Dosages of Concerta® will be defined according to the Swiss Compendium (from 18 to 72 mg/d).
  The psychiatrist will start with the smallest dosage (18 mg) and will adapt it on a weekly basis or on need, depending on tolerance (side effects measured at each visit), clinical response (subjective improvement felt by the patient in terms of attention, impulsivity, and hyperactivity), and according to the observations made by the professionals or patient's entourage in term of attention, impulsivity, hyperactivity, and for this project, behavioral problems. In general, the dose can be increased in 18 mg at weekly intervals.
  The treatment will be monitored weekly the first month, and then monthly, except for side effects which will be monitored daily in prison and every two weeks after release.
  Arms: Pharmaceutical intervention (OROS-MPH)
Drug: Placebo — The placebo will be strictly identical (same packaging, size no. 2 and color according to dosage, with no label).
  Procedure for adjustment of dosage will be the same as in the Concerta arm.
  Arms: Placebo

SUMMARY:
Attention deficit hyperactivity disorder (ADHD) is characterized by difficulties paying attention, poor impulse control, and hyperactive behaviors. It is associated with several health and social detrimental outcomes and leads to increased risks of criminality and recidivism. However, to date, ADHD treatment has been neglected in prison. This project will test the efficacy of ADHD treatment using a randomized controlled trial.

DETAILED DESCRIPTION:
This project aims to compare the efficacy of a three-month in-prison OROS-methylphenidate vs. placebo treatment on the severity of ADHD core symptoms. Secondary outcomes address additional important in-prison and outpatient (in-prison or post-prison) aspects: 1) reduction in acute events in prison (e.g., disciplinary sanctions, violence, misuse of ADHD treatment), 2) evaluation of the risk of recidivism upon release, 3) three-month side effects of treatment, 4) in- and post-prison adherence to medication, 5) in- and post-prison study retention, 6) in- and post-prison costs-benefits of treatment, and 8) one-year rule-breaking behaviour. The outpatient part of the project will highlight long-lasting benefits of a treatment provided during three months while people are detained.

These research questions will be answered using a randomized controlled trial. After randomization, the participants will undertake three months of treatment with OROS-MPH or placebo (1:1 ratio) while they are incarcerated. After three months, all participants will be offered the possibility to have the treatment, but they will remain blinded regarding their initial study group. All of them will benefit of a cognitive-behavioral psycho-education program during detention and a cognitive-behavioral therapy after release.

The RCT will provide empirical-based evidence of the benefits of in-prison ADHD treatment using different perspectives: Clinical, behavioral, rule-breaking-related, and economical. The investigators expect that early detection and treatment of ADHD in prison will be an important public health opportunity and a cost-effective approach, likely to decrease the vulnerability of people living in detention and to promote pathways out criminal involvement.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65
* good command of French
* stay in prison approx. 4 months at eligibility visit
* endorsing clinical diagnostic criteria for DSM-5 ADHD
* providing written informed consent

Exclusion Criteria:

* presence of an acute uncontrolled comorbid psychiatric disorder
* medical contraindication to stimulant prescription
* potential adverse interaction with another medication
* already receive ADHD treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Severity of ADHD core symptoms | 3 months
  Conners Adult ADHD Rating Scale, range 0-78, higher score indicates worse outcome

SECONDARY OUTCOMES:
Number of acute events | 3 months
  Refusal to see doctors, nurses or lawyers, hunger strikes, self-harm events requiring a visit to the medical unit, fights requiring a visit to the medical unit, and disciplinary sanctions
Score of risk of recidivism | 3 months
  Dynamic risk assessment tool will be used to evaluate the risk of recidivism, score 0-30, higher score indicates better outcome
Percentage of adherence to medication | 3 months and 12 months in outpatient care
  Binary variable (yes=adherence to medication, no=absence of adherence to medication)
Percentage of retention to study | 12 months in outpatient care
  Binary variable (yes=remain in the study, no=dropout from the study)
Costs | 3 months (medical and prison-related costs) and 12 months in outpatient care (prison-related costs)
  Medical costs (costs of medical services used by patients (outpatient, emergency, and inpatient resources) and prison-related costs (disciplinary sanctions, use of resources in the prison and in prison staff and recidivism-related costs, average cost for one day in prison), two quantitative variables in Swiss francs.
Number of rule-breaking events | 12 months in outpatient care
  Composite outcome with sanctions recorded in prison and recidivism from the official Swiss criminal records (Federal Office of Statistics, Criminal Conviction Statistics) after release, binary variable (yes=rule-breaking behaviour, no=no rule-breaking behaviour)

OTHER OUTCOMES:
Number of side effects | 3 months
  Side effects according to the Swiss compendium (number of side effects)

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Baggio S, Billieux J, Dirkzwager A, Iglesias K, Moschetti K, Perroud N, Schneider M, Vernaz N, Wolff H, Heller P. Protocol of a monocentric, double-blind, randomized, superiority, controlled trial evaluating the effect of in-prison OROS-methylphenidate vs. placebo treatment in detained people with attention-deficit hyperactivity disorder (BATIR). Trials. 2024 Jan 4;25(1):23. doi: 10.1186/s13063-023-07827-7. PMID 38178233